CLINICAL TRIAL: NCT05097053
Title: A Parallel Group, Prospective, Randomized, Two-arm, Open-label Study to Evaluate the Immunogenicity, Safety, and Tolerability of Heterologous 3rd Boost of MVC-COV1901 in Adults With 2 Doses of ChAdOx1-nCov-19 in 3 Months and 6 Months
Brief Title: A Heterologous 3rd COVID-19 Vaccine of MVC-COV1901 to Evaluate Immunogenicity and Safety in Adults With ChAdOx1-nCov-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taoyuan General Hospital (Other Government)
Collaborators: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TYGH110044
Record Dates: First submitted 2021-10-17; First posted 2021-10-27 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Vaccine
Keywords: COVID-19 Vaccine
MeSH Terms: interventions — MVC-COV1901 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVC-COV1901 vaccine (3-month Interval) (Experimental): There will be approximately 100 participants (Group A) who had received 2 doses of ChAdOx1-nCov-19 and will be vaccinated with MVC-COV1901 at Day 1
  Interventions: Biological: MVC-COV1901(3 Months)
- MVC-COV1901 vaccine (6-month Interval) (Experimental): There will be approximately 100 participants (Group B) who had received 2 doses of ChAdOx1-nCov-19 and will be vaccinated with MVC-COV1901 at Day 85.
  Interventions: Biological: MVC-COV1901(6 Months)

INTERVENTIONS:
Biological: MVC-COV1901(3 Months) — MVC-COV1901 vaccine after a 3-month Interval
  Arms: MVC-COV1901 vaccine (3-month Interval)
Biological: MVC-COV1901(6 Months) — MVC-COV1901 vaccine after a 6-month Interval
  Arms: MVC-COV1901 vaccine (6-month Interval)

SUMMARY:
This primary objective of the study is to measure the anti-SARS-CoV-2 neutralizing antibody titers in adult participants in order to demonstrate the immunogenicity and safety of heterologous third-boost with MVC-COV1901, in terms of the neutralizing antibody GMTs at 28 days after the study intervention. This study also assesses the safety and tolerability of the study intervention and explores the immunogenicity by the antigen-specific immunoglobulin as well as the potential efficacy of study intervention in preventing COVID-19. This study is aimed to recruit participants at single study site in Northern Taiwan.

DETAILED DESCRIPTION:
This a parallel group, prospective, randomized, two-arm, open-label, single-center study to be conducted in approximately 200 healthy participants aged 20 to 64 years who have had their two doses of ChAdOx1-nCov-19 (Astra Zeneca). Preparation and administration of study intervention will be performed by authorized unblinded site personnel. Eligible participants will receive MVC-COV1901 vaccine after a 3-month (Group A: < 16 weeks and ≥ 12 weeks) or 6-month (Group B: < 28 weeks and ≥ 24 weeks) interval apart from their second dose of ChAdOx1-nCov-19.

The study consists of 6 on-site visits:

* Day -28 to Day 1, Visit 1 (Screening)
* Day 1, Visit 2 (study intervention) : randomization Group A and B

Group A:

* Day 1, Visit 2: treatment
* Day 29 ± 3 days, Visit 3
* Day 85 ± 3 days, Visit 4
* Day 169 ± 3 days, Visit 5

Group B:

* Day 1, Visit 2
* Day 85 ± 3 days, Visit 3: treatment
* Day 113 ± 3 days, Visit 4
* Day 169 ± 3 days, Visit 5

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged 20 to 64 years at randomization.
2. Has received two doses of the ChAdOx1-nCov-19 (Astra-Zeneca) 12 to 16 weeks before randomization.
3. Female participant must:

   1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following the last administration of study intervention. Acceptable forms include:

   i.Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii.Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository c.Have a negative pregnancy test
4. Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
5. Participant or the participant's legal representative must understand the procedures of the study and provide written informed consent.

Exclusion Criteria:

1. Pregnant or breast feeding or have plan to become pregnant within 30 days after the last administration of study intervention.
2. Currently receiving or received any investigational intervention within 30 days prior to the first dose of study intervention.
3. Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live-attenuated vaccines within 7 days prior to the first dose of study intervention.
4. Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the first dose of study intervention.
5. Currently receiving or anticipate to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the first dose of study intervention.
6. Currently receiving or anticipate to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks prior to the first dose of study intervention.
7. Major surgery or any radiation therapy within 12 weeks prior to the first dose of study intervention.
8. Has received any other investigational or licensed COVID-19 vaccine.
9. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
10. A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
11. Bleeding disorder considered a contraindication to IM injection or phlebotomy.
12. Known SARS-CoV-2 infection in the recent 3 months prior to the first dose of study intervention.
13. A history of cerebral venous sinus thrombosis, heparin-induced thrombocytopenia or antiphospholipid syndrome.
14. Participant who, in the investigator's judgement, is not in a stable condition and by participating in the study could adversely affect the safety of the participant, interfere with adherence to study requirements or evaluation of any study endpoint. This may include a participant with ongoing acute diseases, severe infections, autoimmune disease, laboratory abnormality or serious medical conditions in the following systems: cardiovascular, pulmonary, hepatic, neurologic, metabolic, renal, or psychiatric.
15. A history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the MVC-COV1901.
16. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the first dose of study intervention.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Primary Immunogenicity | Day1 to 28 days after vaccination
  To evaluate the immunogenicity of heterologous third-boost (MVC-COV1901) in 3 months, compared to 6 months, in terms of neutralizing antibody
  Geometric Mean Titers (GMT)
Primary Safety | Day1 to 28 days after vaccination
  To evaluate the safety and tolerability of heterologous third-boost (MVC-COV1901) from Day 1 to 28 days after the study intervention
  The number and percentage of participants with the occurrence of:
  * Solicited local adverse events (AEs)
  * Solicited systemic AEs
  * Unsolicited AEs

SECONDARY OUTCOMES:
Secondary Immunogenicity | Day 1 and Day 169
  To evaluate the immunogenicity of heterologous third-boost (MVC-COV1901) in terms of antigen-specific immunoglobulin titers
  GMT
Secondary Safety | Day 1 to Day169
  To evaluate the safety of heterologous third-boost (MVC-COV1901), over the study period
  The number and percentage of participants with the occurrence of:
  * MAAEs
  * AESIs
  * VAED
  * SAEs

OTHER OUTCOMES:
Exploratory Efficacy | Day 1 to Day 169
  To estimate the efficacy of heterologous third-boost (MVC COV1901), in the prevention of COVID-19
  * Number of laboratory-confirmed COVID-19 cases occurring ≥ 7 days after study intervention.
  * Number of laboratory-confirmed COVID-19 severe cases occurring ≥ 7 days after study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Yu Cheng, MD.PhD., Principal Investigator — Taoyuan General Hospital
Locations (1):
- Taoyuan General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No